CLINICAL TRIAL: NCT00375414
Title: New Introducer PEG-Gastropexy Does Not Need Prophylactic Antibiotics: Prospective Randomised Double Blind Placebo Controlled Trial
Brief Title: Role of Prophylactic Antibiotics in New Introducer PEG-Gastropexy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Collaborators: Bethanien Krankenhaus gGmbH (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Gastropexy
Record Dates: First submitted 2006-09-12; First posted 2006-09-13 (Estimated); Last update posted 2007-05-07 (Estimated); Status verified 2007-05

CONDITIONS: Head and Neck Neoplasms; Wound Infection
Keywords: Enteral tube feeding,; endoscopic gastropexy,; percutaneous endoscopic gastrostomy,; PEG
MeSH Terms: conditions — Head and Neck Neoplasms; Wound Infection

INTERVENTIONS:
Procedure: PEG-Gastropexy

SUMMARY:
Peristomal infections are the commonest complications of PEG despite prophylactic antibiotics which may result in emergence of resistant micro-organisms like Methicillin resistant Staphylococcus aureus (MRSA). Introducer PEG technique avoids the sojourn of PEG catheter through the oropharynx so chances of infectious complications are negligible. It was not popular because of associated risks and complications. However the new introducer PEG gastropexy has been recently proved to be safe. To determine the incidence of peristomal wound infections during the immediate 7 day post procedure follow up period after the new introducer PEG gastropexy

DETAILED DESCRIPTION:
BACKGROUND:PEG can be performed by pull, push or introducer technique, pull method is the one most commonly used worldwide. PEG site infection is clearly the commonest procedure related complication of PEG placement and the routinely used pull technique has been shown to have quite high (4-30%), peristomal infectious complications. To curtail these infectious complications various gastroenterological societies have recommended giving intravenous prophylactic antibiotics 30 minutes prior to the procedure which has been shown to significantly reduce this complication. Despite this the incidence of peristomal infectious complications remains high post PEG. Another problem associated with the administration of prophylactic antibiotics is the emergence of resistant micro-organisms especially the Methicillin resistant Staphylococcus aureus (MRSA) at the PEG site. Introducer PEG is the technique of PEG placement which avoids the transit of PEG catheter through the oropharynx. Despite its introduction since 19 years back it has not become popular among endoscopists because of technical difficulties and complications associated with it. However the newer introducer PEG technique using endoscopic gastropexy has been shown to be quite safe and easy to perform in recent studies. We at our institute have been performing this procedure since January 2003 and on prospective follow up have found much lower incidence of peristomal infections with it. Recently Maetani et al have already demonstrated in a prospective randomised trial that the introducer type PEG results in fewer infectious complications as compared to conventional pull PEG. There is no study comparing introducer PEG technique with or without administration of prophylactic antibiotics. As in principal, the chances of infections are much lower in the introducer technique. We want to address this issue in a randomised double blind placebo controlled settings in those patients who will as it is unfit to undergo routine pull PEG because of upper gastrointestinal (UGI) malignant stenoses.

SUMMARY: Peristomal infections are the commonest complications of PEG despite prophylactic antibiotics which may result in emergence of resistant micro-organisms like Methicillin resistant Staphylococcus aureus (MRSA). Introducer PEG technique avoids the travel of PEG catheter through the oropharynx which is richly inhabitated with microorganisms so chances of infectious complications at the raw PEG wound are negligible. This technique was not popular because of associated risks and complications in the past which has shown it to result in complications like deflation of balloons, catheter dislodgement, leading to peritonitis etc. However the new introducer PEG gastropexy has been recently proved to be safe. At our institute about 200 PEG procedures are performed annually, out of these 10-12% have tight stenotic stricture in which pull PEG is not possible without dilatation of oropharyngeal tract. We plan to randomise these patients in to 2 groups with and without antibiotics (placebo). PEG will be done using the new introducer PEG, Freka® Pexact CH/FR 15 (Fresenius Kabi, Germany), in which the gastric wall is sutured non surgically to the anterior abdominal wall using 2 silk sutures. Peristomal wound would be assessed daily for 7 days using 2 types of point scores systems (given by Jain and by Gossner) by 2 members of nutrition support team independently. As these are the objective scoring systems, we intend to determine the grades of post procedure peristomal infections in these patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients having very tight stenotic malignant lesions of the upper GI tract (i.e. esophagus and or oropharynx) in whom routine pull PEG is not possible without dilatation/bougeinage of the UGI tract. The GI lumen in patients included in this study would have just sufficiently enough diameters to allow only the passage of thin (8.8 mm) endoscope.

Exclusion Criteria:

* Allergies to Ceftriaxone antibiotics,
* Patients receiving systemic antibiotics,
* Any contraindications to PEG like, severe coagulation disorders, peritonitis, peritoneal carcinomatosis, burns or inability to achieve transillumination.

Ages: 16 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2003-10; Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
peristomal infection rate over a period of 7 days after PEG-gastropexy | cross sectional

CONTACTS AND LOCATIONS:
Overall Officials: Yogesh M Shastri, MD, DNB, Principal Investigator — JW Goethe University Hospital, Frankfurt
Locations (1):
- Department of Medicine I, Division of Gastroenterology and Clinical Nutrition, Johann Wolfgang Goethe-University Hospital,, Frankfurt am Main, Germany

REFERENCES:
- [Derived] Shastri YM, Hoepffner N, Tessmer A, Ackermann H, Schroeder O, Stein J. New introducer PEG gastropexy does not require prophylactic antibiotics: multicenter prospective randomized double-blind placebo-controlled study. Gastrointest Endosc. 2008 Apr;67(4):620-8. doi: 10.1016/j.gie.2007.10.044. PMID 18374024